CLINICAL TRIAL: NCT03352076
Title: A Comparative, Open-Label, Randomized, Parallel Group Study to Determine Intraperitoneal Fluids, Tissue, and Serum Concentrations of VML-0501 Following Five Days of Daily Vaginal Applications of Single Dose of VML-0501 (100 mg Danazol), in Comparison to Five Days of Danazol Treatment Administered as an Oral Capsules (Danatrol) at a Daily Dose of 600 mg, in Two Groups of Twelve Each Consisting of Women With Suspected or Confirmed Endometriosis and Scheduled for Laparoscopy
Brief Title: Study to Determine Intraperitoneal,Tissue, Serum Concentrations of VML-0501 Following Five Days of Daily Vaginal Single Dose of VML-0501 (100 mg Danazol), in Comparison to Oral Danazol Capsules Daily 600 mg), in Women With Signs and Symptoms of Endometriosis Undergoing Laparoscopy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Viramal Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VML-0501-001
Record Dates: First submitted 2017-11-17; First posted 2017-11-24 (Actual); Last update posted 2020-06-12 (Actual); Status verified 2020-06

CONDITIONS: Endometriosis
Keywords: Danazol
MeSH Terms: conditions — Endometriosis | interventions — Danazol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oral Danatrol (Active Comparator): 200 mg orally TDS (600 mg daily) for 5-7 days
  Interventions: Drug: Oral Danatrol
- Vaginal Danazol (Experimental): 100 mg of Danazol Cream to be applied vaginally for 5-7 days on a single daily dose
  Interventions: Drug: Vaginal Danazol

INTERVENTIONS:
Drug: Vaginal Danazol — Proof of mechanism study to establish intraperitoneal and serum concentrations of Danazol
  Arms: Vaginal Danazol
Drug: Oral Danatrol — Proof of mechanism study to establish intraperitoneal and serum concentrations of Danazol
  Arms: Oral Danatrol

SUMMARY:
A Comparative, Open-Label, Randomized, Parallel Group Study to determine Intraperitoneal fluids, tissue, and serum concentrations of VML-0501 following five days of daily vaginal applications of single dose of VML-0501 (100 mg Danazol), in comparison to five days of Danazol treatment administered as an oral capsule (Danatrol) at a daily dose of 600 mg, in two groups of twelve each consisting of women with suspected or confirmed endometriosis and scheduled for laparoscopy.

ELIGIBILITY:
Inclusion Criteria:

* Provide written (personally signed and dated) informed consent before completing any study-related procedure, which means any assessment or evaluation that would not have formed a part of her normal medical care.
* Be a female who has or is suspected to have endometriosis
* Greater than or equal to 18 years of age and less than 42years.
* Scheduled to undergo laparoscopy.
* According to the local practice the women should sign a specific clause on avoiding pregnancy based on the use of two effective methods for birth control (condom and spermicidal) following 30 days after the last dose/application.
* Be non-pregnant undergoing laparoscopy for confirmed or suspected endometriosis within first 10 days of her cycle.
* Have a body mass index (BMI) < 32 kg/m2

Exclusion Criteria:

If any of the following criteria apply, the subject MUST NOT be admitted/continue the study trial.

The subject:

* Is pregnant (if positive-Urine pregnancy test at screening) or lactating;
* Has evidence of drug or alcohol abuse.
* Have used hormonal replacement therapy or Danazol therapy within the past 8 weeks before study entry
* Has any of the following: Epileptic Seizure, Migraine Headache, Angina, Chronic Heart Failure, Obstruction of a Blood Vessel by a Blood Clot, Liver Problems, Kidney Disease, Pregnancy, Combined High Blood Cholesterol and Triglyceride Level, Porphyria
* Undiagnosed abnormal genital bleeding
* Androgen dependant tumour
* Is Allergic to anabolic androgenic steroid.
* Smoker.

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2017-12-28 (Actual); Primary Completion 2019-10-24 (Actual); Study Completion 2020-05-26 (Actual)

PRIMARY OUTCOMES:
Danazol concentration | 6 months
  Concentration in serum and peritoneal fluid

SECONDARY OUTCOMES:
Danazol concentration | 6 months
  Concentration in endometrial tissue found outside the uterus

OTHER OUTCOMES:
Danazol concentration | 6 months
  Concentration in endometrium tissue
Danazol concentration | 6 months
  Concentration in myometrium tissue

CONTACTS AND LOCATIONS:
Overall Officials: Simona Fiore, Dr, Study Director — Viramal Limited
Locations (1):
- Ospedale L. Sacco - Milan-Obgyn Unit, Milan, Italy

IPD SHARING:
Plan to Share IPD: No